CLINICAL TRIAL: NCT00846014
Title: Asthma Exacerbation and Helium-3 MRI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Subjects which fit the strict inclusion criteria were not found.
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Mitchell Albert, Director of Advanced MRI Center, UMASS Medical Sch, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Docket # 12937
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Asthma Exacerbation
Keywords: asthma; exacerbation; Helium; MRI; Lung imaging
MeSH Terms: conditions — Asthma | interventions — Helium-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Asthmatics (Experimental): All subjects will be asthmatics that have had an exacerbation (asthma attack) no more than 48 hours before the imaging session.
  Interventions: Drug: Helium-3

INTERVENTIONS:
Drug: Helium-3 — Patients will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of Helium-3 gas and 667mL of Nitrogen. The first three bags will be administered with a break between each of five to ten minutes. Then the drug aformoterol will be administered and an hour will pass. Then three additional bags will be administered, again with five to ten minutes between each bag.
  Other Names: Hyperpolarized Helium-3

SUMMARY:
The goal of this research is to use Helium-3 MRI to see the changes in airflow of the lungs at different times of an attack. These three stages are immediately after the attack, 1 month later and 4-6 months later.

DETAILED DESCRIPTION:
Asthma is a pulmonary disorder that affects millions of people each year. The exact method of exacerbation is still under some discussion. Currently there is no cure for the disorder but treatment is of a wide variety.

This study is meant to image the asthmatic lung at various time points post exacerbation. Since pulmonary imaging is currently limited to radiation techniques, this method will allow exacerbated images without the unnecessary exposure to radiation.

ELIGIBILITY:
Inclusion Criteria

* At least 18 years old
* Able to speak and read English
* Acute asthma exacerbation, defined as requirement for hospitalization or emergent outpatient visit, and treatment with high dose corticosteroids ( 40mg prednisone or equivalent)
* FEV1 < 80% predicted on the day of MRI
* Attending physician agrees that patient is safe to participate on the day of the MRI scan

Exclusion Criteria

* Evidence of pneumonia, based on chest radiograph obtained within 24 hours of enrollment (if performed)
* Documented fever or requirement for antibiotics
* Unable to hold breath for 10 seconds
* Active smoker or history of at least 10 pack years cigarette smoking
* Chest radiograph with active pulmonary disease, except for changes expected with asthma (hyperinflation, subsegmental atelectasis)
* Admission to ICU
* For inpatients: contraindication to leaving hospital room for MRI as determined by Attending physician and RN on day of MRI
* Any other concurrent active pulmonary disease or other unstable or active medical condition (including suspected active coronary ischemia, acute bleeding), as determined by Attending physician
* Pregnancy as self reported
* Need for cardiac monitoring
* Need supplemental oxygen at an amount of 4L/min or a facemask

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Image and quantify variation in asthmatic lungs at 0, 6 months, and 12 months | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Albert, Ph.D., Principal Investigator — UMASS Medical School
Locations (1):
- UMASS Medical School Advanced MRI Center, Worcester, Massachusetts, United States